CLINICAL TRIAL: NCT06943521
Title: A Phase I/II, Dose-escalation and Dose-optimization Study to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of MT-4561 in Patients With Various Advanced Solid Tumors and to Evaluate Effect of MT-4561 on Pharmacokinetics of Oral Midazolam
Brief Title: A Study of MT-4561 in Patients With Various Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-4561-Z-101
Record Dates: First submitted 2025-03-28; First posted 2025-04-24 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC); Non-small Cell Lung Cancer (NSCLC); Esophageal Cancer; Gastric Cancer; Biliary Tract Cancer; Pancreatic Ductal Adenocarcinoma (PDAC); Breast Cancer; Ovarian Cancer; Cervical Cancer; Endometrial Cancer; Prostate Cancer; Urothelial Carcinoma; Neuroendocrine Tumor (NET); Neuroendocrine Carcinoma (NEC); Soft Tissue Sarcoma; Nuclear Protein in Testis (NUT) Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms; Stomach Neoplasms; Biliary Tract Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Prostatic Neoplasms; Carcinoma, Transitional Cell; Neuroendocrine Tumors; Carcinoma, Neuroendocrine; Sarcoma; Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part 1 (Dose-escalation) (Experimental): Intravenous (IV) infusion of MT-4561 once every week in 28-day cycle, until disease progression or discontinuation criteria are met.
  Interventions: Drug: MT-4561

INTERVENTIONS:
Drug: MT-4561 — i.v.

SUMMARY:
This is a First In Human (FIH), multicenter, open-label, Phase I/II study to evaluate safety, tolerability, Pharmacokinetics (PK), pharmacodynamics, and efficacy of MT-4561 in patients with advanced solid tumors. This study will be conducted in 3 parts.

Part 1 is aimed at evaluating safety, tolerability, PK and pharmacodynamics of MT-4561 and determining the Maximum Tolerated Dose (MTD) using the Bayesian Optimal Interval (BOIN) design.

The study details and doses of Part 2 (dose-optimization) and Part 3 (Drug-Drug Interaction) will be available after review of applicable Part 1 results.

ELIGIBILITY:
Main Inclusion Criteria:

Patients who have failed at least 1 prior therapy and, who have no standard treatment options demonstrated to provide clinical benefit or who are intolerable to or refuse further standard therapies will be enrolled.

* Male or female patient aged 18 years or older at the time of signing the informed consent form
* ≥ 1 measurable lesion by the RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status: 0 to 1
* Life expectancy of at least 3 months
* Adequate bone marrow function
* Adequate hepatic function
* Adequate renal function estimated creatinine clearance ≥ 60 mL/min calculated using the Cockcroft and Gault equation or by institutional method
* Part 1: Patients must have a confirmed histologic or cytologic diagnosis of one of the following solid tumors for participation in the study: head and neck squamous cell carcinoma (HNSCC), non-small cell lung cancer (NSCLC), esophageal cancer, gastric cancer, biliary tract cancer, pancreatic ductal adenocarcinoma (PDAC), breast cancer, ovarian cancer, cervical cancer, endometrial cancer, prostate cancer, urothelial carcinoma, neuroendocrine tumor (NET) or neuroendocrine carcinoma (NEC), soft tissue sarcoma, and NUT carcinoma.

Main Exclusion Criteria:

* Patients with active brain or leptomeningeal metastases
* Any unresolved toxicity ≥ Grade 2 from previous anticancer therapy except for alopecia
* Prior systemic anticancer therapy within 4 weeks before first dose of investigational medicinal product (IMP) or 5 half-lives, whichever is shorter, and prior radiotherapy within 2 weeks before first dose of IMP
* History of congenital long QT syndrome or clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation or Torsades de pointes)
* Patients who received drugs with a known risk of QT interval prolongation or Torsades de pointes within 14 days or 5 half-lives, whichever is shorter, before the start of IMP administration
* QT interval corrected for heart rate using Fridericia's correction (QTcF) > 470 msec at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Event, Dose limiting toxicities (DLTs) | a 28-day cycle
  Part 1 Frequency, duration, and severity (Common Terminology Criteria for Adverse Events [CTCAE] v5.0) of adverse events, dose limiting toxicity (DLT), physical examinations, changes in clinical laboratory values (e.g., hematology, chemistry, and urinalysis), vital signs (e.g., heart rate, blood pressure, respiratory rate), electrocardiogram
  DLTs are defined as any event meeting the DLT criteria at least possibly related to MT-4561 for Cycle 1 (i.e., DLT monitoring window is approximately 28 days). Events with a clear alternative explanation will not be considered DLTs.
Number of Patients with Adverse events (AEs) | Screening through 30 days after last dose
  Part 1 Frequency, duration, and severity (Common Terminology Criteria for Adverse Events [CTCAE] v5.0) of adverse events, dose limiting toxicity (DLT), physical examinations, changes in clinical laboratory values (e.g., hematology, chemistry, and urinalysis), vital signs (e.g., heart rate, blood pressure, respiratory rate), electrocardiogram
  Adverse event: An AE is defined as any untoward medical occurrence in a clinical study patient administered a pharmaceutical product, and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of an IMP, whether it is considered related to the IMP.

SECONDARY OUTCOMES:
Cmax of MT-4561 | Cycle 1 Day 1 through Cycle 2 Day 22 (each cycle is 28 days)
  To determine the pharmacokinetics(PK) profile of MT-4561
time corresponding to occurrence of Cmax (tmax) | Cycle 1 Day 1 through Cycle 2 Day 22 (each cycle is 28 days)
  To determine the pharmacokinetics(PK) profile of MT-4561
minimum observed plasma concentration (Cmin) | Cycle 1 Day 1 through Cycle 2 Day 22 (each cycle is 28 days)
  To determine the pharmacokinetics(PK) profile of MT-4561
area under the concentration-time curve from zero up to 168 hours post-dose (AUC0-168) | Cycle 1 Day 1 through Cycle 2 Day 22 (each cycle is 28 days)
  To determine the pharmacokinetics(PK) profile of MT-4561
Renal clearance (CL) after the first dose and at steady state | Cycle 1 Day 1 through Cycle 2 Day 22 (each cycle is 28 days)
  To determine the pharmacokinetics(PK) profile of MT-4561
dose proportionality | Cycle 1 Day 1 through Cycle 2 Day 22 (each cycle is 28 days)
  To determine the pharmacokinetics(PK) profile of MT-4561
accumulation ratio | Cycle 1 Day 1 through Cycle 2 Day 22 (each cycle is 28 days)
  To determine the pharmacokinetics(PK) profile of MT-4561
Objective Response Rate (ORR) | From Cycle 1 Day 1 until Progressive Disease/Death/or start of new anticancer therapy, up to approximately 3 years
  ORR defined as the proportion of patients with a best overall response of complete response (CR) and partial response (PR) recorded from start of study intervention until the last objective response documented.
Disease control rate (DCR) | From Cycle 1 Day 1 until Progressive Disease/Death/or start of new anticancer therapy, up to approximately 3 years
  DCR defined as the proportion of patients with a best overall response of complete response (CR), partial response (PR), or stable disease (SD).
Clinical benefit rate (CBR) | From Cycle 1 Day 1 until Progressive Disease/Death/or start of new anticancer therapy, up to approximately 3 years
  CBR defined as the proportion of patients with best overall response of complete response (CR), partial response (PR), or who have had stable disease (SD) for a minimum of 6 months after the first dose of study intervention.
Best overall response (BoR) | From Cycle 1 Day 1 until Progressive Disease/Death/or start of new anticancer therapy, up to approximately 3 years
  BoR defined as the best response in the order of complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) among all overall responses recorded from the start of the study intervention until the last objective response recorded.
Duration of Response (DoR) | From Cycle 1 Day 1 until Progressive Disease/Death/or start of new anticancer therapy, up to approximately 3 years
  Investigator Review according to RECIST v1.1 criteria
Progression-Free Survival (PFS) | From Cycle 1 Day 1 until the first documented objective disease progression or death due to any cause, whichever occurs first, up to approximately 3 years
  Investigator Review according to RECIST v1.1 criteria
Overall Survival (OS) | From Cycle 1 Day 1 until Death, up to approximately 3 years
  Investigator Review according to RECIST v1.1 criteria
Duration of stable disease (SD) | From Cycle 1 Day 1 until Progressive Disease/Death/or start of new anticancer therapy, up to approximately 3 years
  Time from the date of the first dose of the study intervention to the first documented progressive disease (PD).

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (6):
- United States (4):
  - University of Southern California, Los Angeles, California
  - START Midwest, Grand Rapids, Michigan
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Japan (2):
  - National Cancer Center Hospital, Chuo-Ku, Tokyo
  - National Cancer Center Hospital East, City

IPD SHARING:
Plan to Share IPD: No